CLINICAL TRIAL: NCT05138471
Title: Addition of Transcranial Direct Current Stimulation and Transcutaneous Electrical Nerve Stimulation to an Education and Exercise Program in Subjects With Chronic Pain Due to Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JOS-2021-01
Record Dates: First submitted 2021-10-04; First posted 2021-12-01 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-01

CONDITIONS: Osteo Arthritis Knee; Chronic Pain
Keywords: tDCS; transcranial direct current stimulation; knee osteoarthritis; TENS; chronic knee pain
MeSH Terms: conditions — Chronic Pain; Osteoarthritis, Knee | interventions — Transcranial Direct Current Stimulation; Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS Active vs TENS Active (Experimental)
  Interventions: Device: transcranial direct current stimulation (tDCS); Device: TENS; Behavioral: Exercise and General Education
- tDCS Active vs TENS Placebo (Experimental)
  Interventions: Device: transcranial direct current stimulation (tDCS); Behavioral: Exercise and General Education
- tDCS Placebo vs TENS Placebo (Placebo Comparator)
  Interventions: Behavioral: Exercise and General Education

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS intervention will consist in placing two electrodes, the cathode on the supraorbital surface on the same side as the painful knee, and the anode on the parietal area, corresponding to the area of the primary motor cortex, on the opposite side. The intensity will be 2 milli amperes (mA) and stimulation will be 20 minutes. The placebo will generate an initial sensation, and then descend until the stimulation is turned off.
  Arms: tDCS Active vs TENS Active; tDCS Active vs TENS Placebo
Device: TENS — TENS intervention will consist in placing two electrodes on the sides of the patella of the affected knee. The frequency will be 10Herzts and the intensity will remain at a sensitive threshold level, without reaching the motor. The placebo will generate a sensation of current to descend to the minimum value that the equipment allows. Stimulation will last for 20 minutes.
  Arms: tDCS Active vs TENS Active
Behavioral: Exercise and General Education — The General Education Intervention consisting in an educational program will be applied to all groups using audiovisual material to increase the subject's knowledge about his/her pathology, about chronic pain and recommendations for supervised exercise based on the NEMEX protocol for osteoarthritis (Ageberg et al.)18: the participants will be taught analytical strengthening exercises (quadriceps and hamstrings) and neuromuscular functional exercises (getting up from the chair or going up a step), with their detailed dosage (2 to 3 series with 10 to 15 repetitions) and a home follow-up model where the participant must record compliance with exercise as well as pain during activity.

SUMMARY:
Knee osteoarthritis has a very high prevalence in the population over 50 years of age. Patients with osteoarthritis often suffer from chronic pain that becomes disabling, affecting both quality of life and mental and physical health. This pathology has also been linked to maladaptive plasticity in the brain, which can contribute to chronic pain. Therapies with neuromodulatory approaches, such as transcranial direct current stimulation (tDCS) and peripheral electrical stimulation (TENS), have been used therapeutically to counteract the maladaptive plasticity of the brain.

Transcranial therapy and TENS can be a possible effective treatment in the rehabilitation services of the health system for the improvement of chronic pain and quality of life in different pathologies, such as chronic low back pain, fibromyalgia or knee and hip osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Adults over fifty years of age with a diagnosis of knee osteoarthritis by radiography.
* Chronic pain of more than six months, compliance with the diagnostic criteria for knee osteoarthritis according to the Osteoarthritis Research Society International (OARSI) guideline:
* Pain in Analog Visual Scale more than 4/10
* Matutinal less than 30 minutes
* Absence of hyperthermia upon palpation in the joint
* Alteration of the bone image
* Crepitus

Exclusion Criteria:

* Patients who can provide low-quality or biased information discriminated by the Mini-Mental State Examination (Score less than 24).
* Severe hearing, visual or sensory impairment or comorbidities that prevent the correct completion of the questionnaires and mobility activities.
* Patients who have undergone knee replacement surgery on the contralateral knee.
* Patients who have received intervention (infiltration, blockages, etc...) in the last 6 weeks.
* Pain due to tendinopathy, knee fracture, low back pain radiating to the knee, or fibromyalgia.
* Patients who decline to participate out of fear or denial of therapy.
* Severe heart disease that prevent exercise.
* Body Mass Index above 45.
* Patients with neuropsychiatric disorders (schizophrenia, epilepsy or bipolar disorders) or taking medication for these conditions (antiepileptic drugs).
* Patients with metallic implants in the area (skull or knee).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Chronic Knee Pain | Through study completion, an average of 1 year.
  The Visual Analogic Scale will be used to assess the impact on chronic knee pain. The values range from 0 to 10 (0 = No pain, 10 = the worst pain).

SECONDARY OUTCOMES:
Function and Quality of Life | Through study completion, an average of 1 year.
  The Western Ontario and McMaster (WOMAC) scale will be used to assess pain, function, and quality of life in knee osteoarthritis and range from 0 to 96 (higher score, worst outcome).
Force | Through study completion, an average of 1 year.
  Using a dynamometer for quadriceps muscle (measurement in Kg, higher score means better outcome).
Balance | Through study completion, an average of 1 year.
  A short physical performance battery (SPPB) will be used to measure balance. SPPB ranges from 0 (worst) to 12 (best).
Gait properties. | Through study completion, an average of 1 year.
  6 Minutes Walk Test (meters) measure exercise tolerance, less than 350 meters is high risk of death in some patients. More meters, more score.
Coordination and Balance | Through study completion, an average of 1 year.
  Timed Up and Go Test (TUG), less than 10 seconds (low risk of falls) more than 20 seconds (high risk of falls).
Uncertainly | Through study completion, an average of 1 year.
  Mishel's Uncertainly Scale (MUIS) range from 55 to 121 (more score, greater uncertainly, worst outcome).
Catastrophizing | Through study completion, an average of 1 year.
  The Pain Catastrophizing Scale (PCS) range from 0 to 52 (more score, greater catastrophizing, worst outcome).
Kinesiophobia | Through study completion, an average of 1 year.
  The Tampa Scale of Kinesiophobia (TSK) range from 11 to 44 (higher values are worst outcome).
Central Sensitization | Through study completion, an average of 1 year.
  8Central Sensitization Inventory (CSI) range from 0 to 100 (higher values are worst outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquina JM Montilla, PhD, PT, Study Director — Director; Mariano MG Gacto, PhD, PT, Study Director — Co-Director
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided